CLINICAL TRIAL: NCT03112811
Title: Influence of Techniques of Chest Physiotherapy on the Respiratory Status and the Hemodynamic Impact in the Pediatric Intensive Care
Brief Title: Influence of Techniques of Chest Physiotherapy in the Pediatric Intensive Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Atelectasis001
Record Dates: First submitted 2017-04-03; First posted 2017-04-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Atelectasis
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intubated infant (Experimental)
  Interventions: Device: Autogenic drainage; Device: Intrapulmonary percussive ventilation
- Extubated infant (Experimental)
  Interventions: Device: Autogenic drainage; Device: Intrapulmonary percussive ventilation

INTERVENTIONS:
Device: Autogenic drainage — The manual technique of the chest physiotherapy to move the secretions
Device: Intrapulmonary percussive ventilation — The instrumental technique of the chest physiotherapy to move the secretions

SUMMARY:
The purpose of this study is to compare the effect of the autogenic drainage and the intrapulmonary percussive ventilation on the levying of the lung atelectasis, by means of the thoracic imaging (thoracic ultrasound and radiography), at the intubated or extubated child with the ventilatory support.

ELIGIBILITY:
Inclusion Criteria:

* Child < 10 kg
* Hospitalization in the pediatric intensive care
* Presence of an atelectasis to the radiography and/or to the lung ultrasound
* Presence of an invasive ventilation or a non-invasive ventilation
* Criteria of cardio-respiratory stability met

Exclusion Criteria:

* Absence of the physiotherapist and the radiologist referents (by ex: at night)
* Prematurity
* Neuromuscular disease
* Ventilation by high-frequency oscillation
* Extraphysical Assistance
* Patient cardiac post-surgery with closure postponed from the thorax. In the closure of the thorax, the patient becomes eligible
* Intracranial pressure > 20 mmHg or clinical signs of intracranial high blood pressure

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2007-04-03 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Atelectasis scores at 20 min | Baseline and at 20 min
  Each atelectasis has a thoracic ultrasound
Change from baseline cardiac frequency at 20 min, 30 min, 50 min, 80 min | Baseline and at 20 min, 30 min, 50 min, 80 min
  Stability of the parameters
Change from baseline respiratory frequency at 20 min, 30 min, 50 min, 80 min | Baseline and at 20 min, 30 min, 50 min, 80 min
  Stability of the parameters
Change from baseline systolic blood pressure at 20 min, 30 min, 50 min, 80 min | Baseline and at 20 min, 30 min, 50 min, 80 min
  Stability of the parameters
Change from baseline diastolic blood pressure at 20 min, 30 min, 50 min, 80 min | Baseline and at 20 min, 30 min, 50 min, 80 min
  Stability of the parameters
Change from baseline oxygen saturation at 20 min, 30 min, 50 min, 80 min | Baseline and at 20 min, 30 min, 50 min, 80 min
  Stability of the parameters
Change from baseline expiratory CO2 at 20 min, 30 min, 50 min, 80 min | Baseline and at 20 min, 30 min, 50 min, 80 min
  Stability of the parameters
Compare the atelectasis scores | Baseline between thoracic ultrasound and chest x-ray
  Compare the atelectasis scores between thoracic ultrasound and chest x-ray

SECONDARY OUTCOMES:
Number of unexpected events | At 20 min
  Pain, desaturation, accidentally extubation

CONTACTS AND LOCATIONS:
Locations (1):
- Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No